CLINICAL TRIAL: NCT00638508
Title: The Analgesic Efficacy of Continuous Infusion of Ketorolac and Ropivacaine at the Wound Site Using ON-Q Pump for Postoperative Pain Management
Brief Title: ON-Q Pump Infusion of Ketorolac and Ropivacaine at the Wound Site for Postoperative Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Collaborators: I-Flow (Industry)
Responsible Party: Principal Investigator, kalpana tyagaraj, Attending, Anesthesiology, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06/07/VA3
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac; Ketorolac Tromethamine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketorolac (Active Comparator): Patients will receive Ketorolac at 5 mg/hr not to exceed 120 mg/day
  Interventions: Drug: Ketorolac
- Ketorolac with Ropivacaine (Experimental): Patients will receive Ketorolac 5 mg and Ropivacaine 0.5% (Group 2) via an infusion catheter at the incision site
  Interventions: Drug: Ketorolac and Ropivacaine

INTERVENTIONS:
Drug: Ketorolac — Patients will receive Ketorolac at 5 mg/hr not to exceed 120 mg/day
  Other Names: Toradol
  Arms: Ketorolac
Drug: Ketorolac and Ropivacaine — Patients will receive Ketorolac at 5 mg/hr plus 0.5% Ropivacaine
  Other Names: Toradol and Naropin
  Arms: Ketorolac with Ropivacaine

SUMMARY:
After surgery it is normal to experience some pain at the site of operation. In order to reduce the pain, medication such as Morphine is injected into a vein using a Patient Controlled Analgesia (PCA) pump that is kept at bed side, and is activated by the patient when needed. However, Morphine is an opioid drug, which can cause side effects such as sedation, nausea, vomiting, and reduced breathing on prolonged use. In addition to the opioid drugs, local anesthetics, and other drugs called Non steroidal anti inflammatory drugs (NSAIDs) have been injected locally to provide prolonged pain relief without the side effects of morphine. Recently a portable device called ON-Q pump has been developed to continuously infuse the local anesthetic through 2 small catheters inserted at the wound site. The ON-Q Pump is a small tennis ball sized unit made of a soft synthetic material that slowly infuses the drug through the catheters by elastic force. This pump is very safe and is attached to a bedside pole or the patient's hospital gown. This pump has already been approved by the FDA for clinical use, and has been reported to provide effective pain management after some surgical procedures.

The primary aim of the present study is to evaluate the relative efficacy of the drugs Ketorolac and Ropivacaine infused through the ON-Q pump in reducing the pain following gynecologic surgery. Ketorolac and Ropivacaine are approved drugs that are frequently used for post operative pain relief. Our hypothesis is that these two drugs in combination will provide better analgesia than Ketorolac alone.

DETAILED DESCRIPTION:
This study would include a total of 60 patients randomized into 2 equal groups. Patients will be interviewed in the holding area and informed signed consent will be obtained. Patients will be induced with general anesthesia in keeping with standard practice. At the end of surgical procedure, before the patient is extubated, the Surgeon will secure the 2 catheters of the ON-Q pump at two levels of the fascia near the incision site. First the surgeon will instill at the wound site a bolus dose of 30 ml of 0.9% saline with 10 mg Ketorolac in Group I, or 30 ml of saline with 0.5% Ropivacaine and 10 mg Ketorolac in Group II patients. Then the continuous infusion with the ON-Q pump will be started at 4 ml/hr, and Group I patients will receive saline with Ketorolac at 5 mg/hr not to exceed 120 mg per day, and Group II will receive saline with 0.5% Ropivacaine plus Ketorolac at 5 mg/hr. Patients will be extubated, as per standard anesthetic practice. All patients will receive anti ulcer medication. On arrival at the Post Anesthesia Care Unit (PACU), the patient will receive an i.v. PCA pump, which will administer Morphine Sulfate 2 mg in incremental doses on demand by the patient.

A blinded investigator will collect the study data from each patient at 6, 12, 24, and 48 hrs postoperative periods. The data collected would include 1) Visual Analog Scale (VAS) scores for pain at rest, on coughing and on moving, 2) PCA demands by the patient and actual deliveries of morphine, 3) "rescue" analgesic requirements (for pain score of 4 or greater). 4) VAS scores for Nausea, drowsiness, and satisfaction, and 5) number of vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patients belonging to ASA class I to II classification who are undergoing abdominal gynecologic surgery will be included in the study.

Exclusion Criteria:

* Patients who are allergic to NSAIDs, Asthmatics, and those who have peptic ulcer, sepsis, or coagulation problems will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana Tyagaraj, M.D., Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac With Rpopivacaine: Patients will receive Ketorolac 5 mg and Ropivacaine 0.5% via an infusion catheter at the incision siteKetorolac and Ropivacaine
Period: Overall Study
Arm/Group | Ketorolac | Ketorolac With Rpopivacaine
Started | 35 | 32
Completed | 30 | 30
Not Completed | 5 | 2
Not completed — Physician Decision | 5 | 2

BASELINE CHARACTERISTICS:
Population: Overall number of participants: 35 in Ketorolac group and 32 in Ketorolac with Ropivacaine group.
  Number of participants analyzed: 30 in each group. 5 participants from the ketorolac and 2 participants from the Ketorolac with Ropivacaine group were omitted from the study.
  Reason for omission- Physician decision.
Groups:
- Ketorolac With Ropivacaine: Patients will receive Ketorolac and Ropivacaine 0.5% via an infusion catheter at the incision site.
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Ketorolac With Ropivacaine | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Full Range); unit: years] — Population: Overall number of participants: 35 in Ketorolac group and 32 in Ketorolac with Ropivacaine group.
  Number of participants analyzed: 30 in each group. 5 participants from the ketorolac and 2 participants from the Ketorolac with Ropivacaine group were omitted from the study.
  Reason for omission- Physician decision.
  years | 25 [18 to 45] | 25 [18 to 45] | 25 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Overall number of participants: 35 in Ketorolac group and 32 in Ketorolac with Ropivacaine group.
  Number of participants analyzed: 30 in each group. 5 participants from the ketorolac and 2 participants from the Ketorolac with Ropivacaine group were omitted from the study.
  Reason for omission- Physician decision.
  Participants
    Female | 30 | 30 | 60
    Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Overall number of participants: 35 in Ketorolac group and 32 in Ketorolac with Ropivacaine group.
  Number of participants analyzed: 30 in each group. 5 participants from the ketorolac and 2 participants from the Ketorolac with Ropivacaine group were omitted from the study.
  Reason for omission- Physician decision.
  Participants
    United States | 30 | 30 | 60
Pain score [Mean (Standard Deviation); unit: units on a scale] — Patients report pain scores using Visual Analog Scale (VAS) . This scale measures the severity of pain and ranges from from 1-10, "1" being minimal pain intensity and "10" being maximal pain intensity. Population: Overall number of participants: 35 in Ketorolac group and 32 in Ketorolac with Ropivacaine group.
  Number of participants analyzed: 30 in each group. 5 participants from the ketorolac and 2 participants from the Ketorolac with Ropivacaine group were omitted from the study.
  Reason for omission- Physician decision.
  units on a scale | 6.7 (2.2) | 6.2 (2.9) | 6.40 (2.6)
Rescue analgesia utilization [Mean (Standard Deviation); unit: milligrams] — Data is obtained regarding use of additional pain medications for breakthrough pain like morphine and acetaminophen with codeine. Rescue analgesics are converted to morphine equivalents and reported in milligrams. Population: Overall number of participants: 35 in Ketorolac group and 32 in Ketorolac with Ropivacaine group.
  Number of participants analyzed: 30 in each group. 5 participants from the ketorolac and 2 participants from the Ketorolac with Ropivacaine group were omitted from the study.
  Reason for omission- Physician decision.
  milligrams | 6.3 (1.9) | 4.0 (2.9) | 5.2 (2.8)
Age [Median (Full Range); unit: years] — Age of the participating patients, reported in years. Population: Overall number of participants: 35 in Ketorolac group and 32 in Ketorolac with Ropivacaine group.
  Number of participants analyzed: 30 in each group. 5 participants from the ketorolac and 2 participants from the Ketorolac with Ropivacaine group were omitted from the study.
  Reason for omission- Physician decision.
  years | 27 [18 to 45] | 26 [18 to 45] | 27 [18 to 45]

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores at Rest
Description: Patients report pain scores at rest using Visual Analog Scale (VAS). This scale measures the severity of pain and ranges from from 1-10, "1" being minimal pain intensity and "10" being maximal pain intensity.
Time Frame: 1 hour after the surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 6.7 (2.2) | 6.2 (2.9)

2. Primary Outcome: Pain Score at Rest
Description: Patients report pain scores at rest using Visual Analog Scale (VAS). This scale measures the severity of pain and ranges from 1-10, "1" being minimal pain intensity and "10" being maximal pain intensity.
Time Frame: At the end of 6 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 3.6 (2.3) | 4.4 (2.5)

3. Primary Outcome: Pain Scores at Rest
Description: Pain scores at rest were measured using the Visual Analog Scale (VAS) at the end of 48 hours. This scale measures the severity of pain and ranges from 1-10, "1" being minimal pain intensity and "10" being maximal pain intensity.
Time Frame: 48 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ketorolac With Ropivacaine: Patients will receive Ketorolac 5 mg/hour and Ropivacaine 0.5% via an infusion catheter at the incision site
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 1.4 (1.6) | 1.6 (2.1)

4. Primary Outcome: Pain Score on Coughing
Description: Pain scores on coughing were measured using the Visual Analog Scale (VAS) at the end of 48 hours. This scale measures the severity of pain and ranges from 1-10, "1" being minimal pain intensity and "10" being maximal pain intensity.
Time Frame: 1 hour after the surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ketorolac With Ropivacaine: Patients will receive Ketorolac and Ropivacaine 0.5% (Group 2) via an infusion catheter at the incision site
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 7.6 (2.2) | 7.5 (2.5)

5. Primary Outcome: Pain Scores on Coughing
Description: Pain scores on coughing were measured using the Visual Analog Scale (VAS) at the end of 6 hours after surgery. This scale measures the severity of pain and ranges from 1-10, "1" being minimal pain intensity and "10" being maximal pain intensity.
Time Frame: 6 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 5.3 (2.5) | 6.2 (2.4)

6. Primary Outcome: Pain Scores on Coughing
Description: Pain scores on coughing were measured using the Visual Analog Scale (VAS). This scale measures the severity of pain and ranges from 1-10, "1" being minimal pain intensity and "10" being maximal pain intensity.
Time Frame: 48 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 3.4 (2.7) | 2.8 (2.3)

7. Primary Outcome: Pain on Movement
Description: Pain scores on movement was assessed using the Visual Analog Scale (VAS). This scale measures the severity of pain and ranges from 1-10, "1" being minimal pain intensity and "10" being maximal pain intensity.
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 7.7 (1.9) | 7.3 (2.9)

8. Primary Outcome: Pain Scores on Movement
Description: Pain scores on movement were assessed using the Visual Analog Scale (VAS) at the end of 6 hours. This scale measures the severity of pain and ranges from 1-10, "1" being minimal pain intensity and "10" being maximal pain intensity.
Time Frame: 6 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 5.7 (2.3) | 26.2 (2.7)

9. Primary Outcome: Pain on Movement
Description: Pain scores on movement were measured 48 hours after surgery using the Visual Analog Scale (VAS). This scale measures the severity of pain and ranges from 1-10, "1" being minimal pain intensity and "10" being maximal pain intensity.
Time Frame: 48 hours afetr surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 3.1 (2.5) | 2.5 (1.9)

10. Secondary Outcome: Morphine Equivalents Utilization
Description: Utilization of morphine and morpine equivalents for rescue analgesia was reviewed and calculated in milligrams.
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: miliigrams
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
miliigrams | 6.3 (1.9) | 4 (2.9)

11. Secondary Outcome: Morphine Equivalents
Description: Utilization of morphine and morphine equivalents for rescue analgesia was reviewed and calculated in milligrams.
Time Frame: 12 hours after surgery
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
milligrams | 2.1 (1.4) | 1.5 (1.1)

12. Secondary Outcome: Morphine Equivalents
Description: Utilization of morphine and morphine equivalents for rescue analgesia, was reviewed and calculated in milligrams.
Time Frame: 48 hours afetr surgery
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
milligrams | 4.2 (2.5) | 4.6 (1.9)

13. Secondary Outcome: DROWSINESS
Description: The severity of drowsiness was measured using Visual Analog Scale (VAS). The VAS scale ranges from 1-10, "1" meaning minimally drowsy and "10" meaning maximally drowsy.
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 4 (2.7) | 4.4 (2.7)

14. Secondary Outcome: DROWSINESS
Description: as for outcome 13
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 0.6 (1.7) | 0.1 (0.4)

15. Secondary Outcome: NAUSEA
Description: The severity of nausea was measured using Visual Analog Scale (VAS). The VAS scale ranges from 1-10, "1" meaning minimally nauseous and "10" meaning maximally nauseous.
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 0.6 (1.6) | 0.9 (2.0)

16. Secondary Outcome: NAUSEA
Description: as for outcome 15
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 0.3 (0.9) | 0.4 (1.8)

17. Secondary Outcome: VOMITING
Description: Data on number of episodes of vomiting was obtained, 6 hours after the surgery. The number of episodes were reported in numerical values, the lower numbers indicating fewer episodes and the higher numbers indicating more number of episodes of vomiting.
Time Frame: 6 hours after surgery
Measure: Mean (Standard Deviation); unit: EPISODES
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
EPISODES | 0.2 (0.6) | 0.1 (0.3)

18. Secondary Outcome: VOMITING
Description: Data on number of episodes of vomiting was obtained, 12 hours after the surgery. The number of episodes were reported in numerical values, the lower numbers indicating fewer episodes and the higher numbers indicating more number of episodes of vomiting.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: EPISODES
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
EPISODES | 0 (0) | 0 (0)

19. Secondary Outcome: PATIENT SATISFACTION
Description: Patient's overall satisfaction was measured using Visual Analog Scale (VAS). This scale ranges from 1-10, "1" indicating least satisfied and "10" indication very well satisfied.
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 5.4 (2.6) | 4.9 (2.8)

20. Secondary Outcome: PATIENT SATISFACTION
Description: as for outcome 19
Time Frame: 48 hours afetr surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ketorolac With Ropivacaine
Number analyzed (Participants) | 30 | 30
units on a scale | 8.5 (1.4) | 8.5 (1.6)

ADVERSE EVENTS:
Time Frame: one year
Groups:
- Ketorolac and Ropivacainr: Patients will receive Ketorolac and Ropivacaine 0.5% via an infusion catheter at the incision site.
Arm/Group | Ketorolac | Ketorolac and Ropivacainr
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No